CLINICAL TRIAL: NCT00553228
Title: Immunization of Women With Diphtheria and Tetanus Toxoids Combined With Acellular Pertussis (Tdap) During the Mid Third Trimester of Pregnancy: An Evaluation of the Potential for Immunological Protection for the Neonate
Brief Title: Pertussis Maternal Immunization Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Scott Halperin (Other)
Collaborators: IWK Health Centre (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Scott Halperin, Dr Scott Halperin, Dalhousie University
Organization: Dalhousie University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAL07-01
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Pregnant Women
Keywords: maternal immunization; whooping cough; pertussis
MeSH Terms: conditions — Whooping Cough | interventions — adacel; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group I (Experimental): Tdap
  Interventions: Biological: Tdap
- group 2 (Active Comparator): Td
  Interventions: Biological: Td

INTERVENTIONS:
Biological: Tdap — 0.5 mL IM once at visit #2
  Other Names: Adacel
  Arms: group I
Biological: Td — 0.5 mL IM once at visit #2
  Other Names: Diphtheria and tetanus toxoids, adsorbed
  Arms: group 2

SUMMARY:
The purpose of this study is to assess whether immunization against pertussis in the mid third trimester of pregnancy provides passive protection to the infant by transfer of IgG transplacentally and by transfer of secretory IgA (and possibly IgG) in breast milk, sufficient to protect the infant against pertussis disease in the critical neonatal period, without suppressing the infant's immune response to active immunization and disease

DETAILED DESCRIPTION:
The purpose of this study is to assess the potential of providing initial immunological protection to the neonate by providing passive placentally transferred serum antibodies and breast milk antibodies against pertussis antigens (PT, FHA, PRN, FIM). This will be accomplished by

* determining the rate of maternal antibody decline from time of immunization until 12 months postpartum by measuring antibody levels in serum, saliva, and breast milk at specified intervals;
* determining levels of antibody transferred to the neonate relative to the interval from immunization to delivery;
* comparing levels of transplacentally transferred antibody with those achieved after the first, second, and third dose of the primary immunization series; and
* determining whether maternal immunization interferes with active antibody production following licensed DTaP-IPV-Hib in infants of women immunized during the mid third trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age and over.
* Women who, at ≥30-<32 weeks gestation, are at low risk for complications as determined by the obstetrical algorithm for identification of eligible subjects and the obstetrical risk assessment form.
* Signed, informed consent.

Exclusion Criteria:

* Failure to meet eligibility criteria as determined by the obstetrical algorithm for identification of eligible subjects and the obstetrical risk assessment form.
* History of significant medical disorder (such as bleeding disorders, cancer, autoimmune disease, immunodeficiency (including HIV-infected individuals, transplant recipients), seizure disorder or significant psychiatric illness, drug or alcohol dependence).
* Receipt of any high-dose daily corticosteroids (inhaled steroids are acceptable) within 2 weeks of study entry. High dose is defined as a dose of ≥20 mg of prednisone daily or equivalent.
* History of physician-diagnosed or laboratory-confirmed pertussis within the past 5 years.
* Personal history (verbal or documented) of ever having received Tdap.
* Personal history (verbal or documented) of having received Td immunization within the past 2 years.
* History of febrile illness (>37.8ºC orally) within the past 72 hours (immunization may be deferred).
* History of sensitivity to any component of Tdap.
* Receipt of blood products or immunoglobulin within 3 months of study entry (except RH-negative women who receive immunoglobulin during pregnancy are eligible).
* Receipt of any vaccines within 2 weeks of study vaccine (except influenza vaccine which may be given concurrently).
* Failure to give written, informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2007-11; Primary Completion 2015-12-09 (Actual); Study Completion 2015-12-09 (Actual)

PRIMARY OUTCOMES:
Comparison of serum IgG antibody levels against PT, FHA, PRN, FIM between Tdap and Td groups | birth, 2, 4, 6, 7, 12, and 13 months of age

SECONDARY OUTCOMES:
Safety of Tdap in pregnancy including pregnancy outcome and developmental assessment. | developmental screening at 1 year of age

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Halperin, MD, Principal Investigator — Dalhousie Univeristy - Canadian Center for Vaccinology
Locations (1):
- Clinical Trial Research Center - Canadian Center for Vaccinology, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Brousseau N, Angers-Goulet ME, Bastien R, Ye L, Sadarangani M, Halperin SA. Vaccination during pregnancy and modulation of IgG response to pertussis vaccines in infants: The impact of different vaccine formulations. Vaccine. 2024 Apr 2;42(9):2138-2143. doi: 10.1016/j.vaccine.2024.03.015. Epub 2024 Mar 8. PMID 38461048
- [Derived] Halperin SA, Langley JM, Ye L, MacKinnon-Cameron D, Elsherif M, Allen VM, Smith B, Halperin BA, McNeil SA, Vanderkooi OG, Dwinnell S, Wilson RD, Tapiero B, Boucher M, Le Saux N, Gruslin A, Vaudry W, Chandra S, Dobson S, Money D. A Randomized Controlled Trial of the Safety and Immunogenicity of Tetanus, Diphtheria, and Acellular Pertussis Vaccine Immunization During Pregnancy and Subsequent Infant Immune Response. Clin Infect Dis. 2018 Sep 14;67(7):1063-1071. doi: 10.1093/cid/ciy244. PMID 30010773
- See also: Canadian Center for Vaccinology Home Page — http://centerforvaccinology.ca